CLINICAL TRIAL: NCT02889471
Title: Routine Nasobiliary Insertion During ERCP to Prevent, Diagnose and Treat of Biliary Injury in High Risk Patients.
Brief Title: Routine Nasobiliary Insertion During ERCP in High Risk Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, MD, Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: fac.med.07
Record Dates: First submitted 2016-08-30; First posted 2016-09-05 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Gallstones Complicated by CBD Stones
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- ERCP with nasobiliary catheter (Experimental)
  Interventions: Procedure: ERCP with NB
- ERCP only (Active Comparator)
  Interventions: Procedure: ERCP alone

INTERVENTIONS:
Procedure: ERCP with NB — ERCP with NB catheter for introperative tans-nasobiliary cholangiography
  Arms: ERCP with nasobiliary catheter
Procedure: ERCP alone — ERCP alone followed with standard laparoscopic cholecystectomy
  Arms: ERCP only

SUMMARY:
110 patients with common bile duct (CBD) stones and had one or more anther preoperative predictors for high risk for difficult cholecystectomy admitted to departement of surgery of Minia university hospital for ERCP then laparoscopic cholecystectomy (LC). the patient divided into 2 equal group. in group 1, nasobiliary (NB) catheter was inserted during ERCP after CBD clearance. In group 2, only CBD clearance was done. In all patients LC was done within the same week of ERCP. Tans-nasobiliary Intraoperative cholangiography was done and methylene blue injected at the end of the procedure to detected any leak in NB group

DETAILED DESCRIPTION:
110 patients with common bile duct (CBD) stones and had one or more anther preoperative predictors for high risk for difficult cholecystectomy as , age > 65 , male sex, obesity, acute cholecystitis, previous upper abdominal surgery, and certain ultrasonographic findings i.e. distended gall bladder (GB), thickened GB wall, pericholecystic fluid collection and impacted stone etc. these patients admitted to department of surgery of Minia university hospital for ERCP followed with laparoscopic cholecystectomy (LC). the patient divided into 2 equal group. in group 1, nasobiliary (NB) catheter was inserted during ERCP to settle high up in the intrahepatic biliary tree after complete CBD clearance. In group 2, only CBD clearance was done. In all patients LC was done within the same week of ERCP. sequential, multiple, step after step, tans-nasobiliary Intraoperative cholangiography was done during every step in cholecystectomy especially during dissection of calot's triangle and just before clipping of supposed cystic duct (CD) to make sure that the structure supposed to be CD was not the CBD. after the end of procedure methylene blue is injected from the the NB to detected any leak and if present

ELIGIBILITY:
Inclusion Criteria:

* patients with GB stone complicated with CBD stones
* accept to share in the study
* the presence of one or more preoperative predictors for high risk for difficult cholecystectomy
* patient fit for LC

Exclusion Criteria:

* patients< 18 and >80
* unfit for surgery
* didn't accept to share in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
biliary injury | 2 weeks
  the incidence of biliary injury complicating cholecystectomy either discovered intraoperative or postoperative
conversion to open | 6 hours
  incidence of conversion to open

SECONDARY OUTCOMES:
operative time | 6 hours
  operative time from skin incision till closure
hospital stay | one month
  time of hospital stay
mortality | one month
  incidence of operative related mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Minya university hospital, Minya, Egypt